CLINICAL TRIAL: NCT02473263
Title: Samu Save Sepsis: Early Goal Directed Therapy in Pre Hospital Care of Patients With Severe Sepsis and/or Septic Shock
Acronym: SSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01030-47
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Severe Septic Syndrome (Severe Sepsis and Septic Shock) Diagnosed and Treated by Mobile Intensive Care Unit
Keywords: Severe septic syndrome; mobile intensive care unit; strategy; antibiotics; hemodynamic optimization
MeSH Terms: conditions — Toxemia; Sepsis; Shock, Septic; Disease | interventions — Ceftriaxone; Piperacillin, Tazobactam Drug Combination; Norepinephrine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (No Intervention): No antibiotic administration and no hemodynamic target are required
- Aggressive (Active Comparator): Antibiotics (Ceftriaxone or piperacillin tazobactam) administration, hemodynamic optimization and opotherapy (norepinephrine, hydrocortisone) when required should be performed in the first 60 minutes after contact with the patient
  Interventions: Drug: Ceftriaxone; Drug: Piperacillin tazobactam; Drug: Norepinephrine; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Ceftriaxone — Ceftriaxone 2g IV will be infused in the first 60 minutes, for non nosocomial severe septic syndrome
  Arms: Aggressive
Drug: Piperacillin tazobactam — Piperacillin/tazobactam 4g IV will be infused in the first 60 minutes, for nosocomial severe septic syndrome
  Arms: Aggressive
Drug: Norepinephrine — Norepinephrine will be infused after failure of hemodynamic optimization using vascular fluid loading
  Arms: Aggressive
Drug: Hydrocortisone — Hydrocortisone 100mg IV will be infused after failure of hemodynamic optimization using norepinephrine with at least 1.5mg/h
  Arms: Aggressive

SUMMARY:
The purpose of this study is to determine whether an aggressive strategy of severe sepsis patients since pre hospital care, including early antibiotics administration, hemodynamic optimization, and opotherapy when indicated, could reduce mortality

DETAILED DESCRIPTION:
Major prognostic factor in sepsis management is rapidity of treatments implementation. In 2001, Rivers observed a reduction in mortality through early hemodynamic optimization. In 2009, Arnold emphasizes that establishing more early antibiotic therapy allowed a further reduction of mortality.

In France, pre hospital care is based on mobile intensive care unit (MICU) called SMUR. SMUR is consisting of a driver, a nurse and an emergency physician.

Actually in France, management of severe septic syndrome (severe sepsis and septic shock) are not standardized and based on a "conventional" strategy at the discretion of the emergency physician. Antibiotics are given in only two cases: fulminans purpura and meningitis. Hemodynamic optimization is not a standard of care and no recommendation exist for hemodynamic targets.

An "aggressive" strategy based on early antibiotics administration, hemodynamic optimization and opotherapy when required could be initiated by SMUR since first contact with the patient before hospital admission.

We assume that an "aggressive" strategy initiated during the first 60 minutes of prehospital stage compared to "conventional" strategy could allow to reduce mortality in severe sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

All patients fulfilling the following criteria:

* Age ≥ 18 years
* Patient with suspected severe infection defined by the existence of a suspected infection AND

  * Hypotension before vascular fluid loading AND/OR
  * Lactataemia greater than 4 mmol/l AND/OR
  * Glasgow scale lower than 13 AND/OR
  * Mottling score greater than 2
* Patient with a septic shock

Exclusion Criteria:

* Age <18 years or Unable
* Pregnant
* Severe concomitant pathology requiring urgent care(i.e.epilepsy)
* Status "not to be reanimated" life expectancy less than 6 months with no indication of reanimation support ( prior decision on care limitation).
* Fulminans purpura
* True allergy to beta-lactam defined by an angioedema or by an anaphylactic shock during a prior exposure to beta-lactam.
* Patient who have already received hemodynamic optimization or antibiotic treatment before the MICU's (Mobile Intensive Care Unit) care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Number of death | 28 days

SECONDARY OUTCOMES:
Number of death | 90 days
Number of death | at hospital discharge time, estimated at 90 days
Number of days of stay in intensive care unit | at Intensive Care Unit discharge time, estimated at 90 days
Number of days of stay at hospital | at hospital discharge time, estimated at 90 days
Number of days of vasopressor support | at Intensive Care Unit discharge time, estimated at 90 days
Number of days of mechanical ventilation support | at Intensive Care Unit discharge time, estimated at 90 days
Number of days of renal replacement therapy | at Intensive Care Unit discharge time, estimated at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, Principal Investigator — Anesthesiology, Intensive Care Unit and emergency department - Necker Hospital - 149 rue de Sèvres 75015 Paris - France
Locations (1):
- Anesthesiology, Intensive Care Unit and emergency department - Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Pottecher T, Calvat S, Dupont H, Durand-Gasselin J, Gerbeaux P; SFAR/SRLF workgroup. Haemodynamic management of severe sepsis: recommendations of the French Intensive Care Societies (SFAR/SRLF) Consensus Conference, 13 October 2005, Paris, France. Crit Care. 2006;10(4):311. doi: 10.1186/cc4965. PMID 16941754
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Intensive Care Med. 2008 Jan;34(1):17-60. doi: 10.1007/s00134-007-0934-2. Epub 2007 Dec 4. PMID 18058085
- [Background] Sebat F, Johnson D, Musthafa AA, Watnik M, Moore S, Henry K, Saari M. A multidisciplinary community hospital program for early and rapid resuscitation of shock in nontrauma patients. Chest. 2005 May;127(5):1729-43. doi: 10.1378/chest.127.5.1729. PMID 15888853